CLINICAL TRIAL: NCT00509197
Title: Should Non-eosinophilic Asthmatic Subjects be Treated With Inhaled Corticosteroids?
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to complete the recruitment.
Sponsor: Université de Montréal (Other)
Collaborators: University of Ottawa (Other); Laval University (Other); University of British Columbia (Other); McGill University (Other); University of Calgary (Other)
Responsible Party: Principal Investigator, Catherine Lemiere, MD,MSc, Université de Montréal
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SFA110717
Record Dates: First submitted 2007-07-27; First posted 2007-07-31 (Estimated); Results first posted 2016-08-15 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-07

CONDITIONS: Asthma
Keywords: Asthma; Non-eosinophilic Asthma; sputum eosinophils; Inhaled Corticosteroids
MeSH Terms: conditions — Asthma | interventions — Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active treatment group (A) (Active Comparator): Intervention : treatment with inhaled corticosteroids (Fluticasone) will be administered to this group
  Interventions: Drug: Fluticasone
- Control group treated with placebo (B) (Placebo Comparator): treatment with placebo
  Interventions: Drug: Placebo (sham inhaler)

INTERVENTIONS:
Drug: Placebo (sham inhaler)
  Other Names: Sham inhaler
  Arms: Control group treated with placebo (B)
Drug: Fluticasone — Fluticasone 250mcg bid for one month
  Other Names: Flovent
  Arms: Active treatment group (A)

SUMMARY:
The efficacy of inhaled corticosteroids (ICS) in asthmatic subjects showing no sputum eosinophils is controversial. The broad aim of this study is to assess whether ICS alone or in combination with long-acting beta-2 agonists are an effective treatment in non-eosinophilic asthmatic subjects. Methods: The investigators will perform a randomized double-blind, placebo-controlled, multicenter study comparing the efficacy of ICS and placebo for 4 weeks followed by a 4-week open treatment period with ICS/salmeterol in steroid-naïve asthmatic subjects without sputum eosinophilia. The primary outcome will be the the Asthma Control Questionnaire (ACQ) score after four weeks of treatment by ICS or placebo.

This study will determine whether or not non-eosinophilic asthmatic subjects respond to ICS and if they further benefit from the addition of a long-acting beta-2 agonists. This study will also determine whether or not the assessment of airway inflammation should be performed in every asthmatic patient in order to give the most appropriate treatment.

DETAILED DESCRIPTION:
General objective: To assess whether inhaled corticosteroids alone or in combination with long-acting beta-2 agonists are an effective treatment in non-eosinophilic asthmatic subjects.

Specific objective 1. To compare the change in clinical and functional outcomes after treatment with fluticasone or placebo in non-eosinophilic asthmatic subjects.

Specific objective 2. To assess whether the combination of inhaled corticosteroids (ICS) and with long-acting beta-2 agonists provides an improvement of asthma control compared to the treatment with ICS or placebo in non-eosinophilic asthmatics.

Hypothesis: Treatment with ICS induces a significant clinical and physiologic improvement of non-eosinophilic asthmatic subjects. ICS/Salmeterol also provides a clinical and physiologic benefit compared to placebo.

Primary end point: Asthma Control Questionnaire (ACQ) score after 4 weeks of treatment with ICS or placebo.

The Asthma Control Questionnaire has been chosen as a primary outcome since it is the most relevant clinical measure to assess asthma control over a short period of time. In patients whose asthma is stable between clinic visits, reliability of the ACQ is high (intraclass correlation coefficient (ICC)=0.90). Furthermore, the questionnaire is also very responsive to changes in asthma control(7). Therefore, this is the ideal tool to assess and compare the changes in asthma control over a short period of time. This instrument has the advantage of including both asthma symptoms as well as forced expiratory flow in one second (FEV1). A change of ACQ of 0.5 has been shown to be clinically significant. Therefore, we will be able to assess whether or not a treatment with ICS has the ability to significantly improve asthma control in non-eosinophilic asthmatic subjects. The questionnaire is provided in appendix III. Other functional and clinical outcomes such as quality of life, FEV1, provocative concentration of methacholine inducing a 20% fall in FEV1 (PC20), number of rescue medication and number of asthma exacerbations will also be assessed as secondary outcomes.

The study has two steps: The first step will be a randomized double-blind, placebo-controlled, multicenter study comparing the efficacy of ICS and placebo for 4 weeks in asthmatic subjects without sputum eosinophilia followed by an open ICS/salmeterol 4-week treatment for all subjects. (See study design in appendix III).

Inclusion criteria One hundred subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Are between 18 and 70 years of age at the time of signing the informed consent.
* Have a diagnosis of asthma according to the Guidelines for the Diagnosis and Management of Asthma and have not been treated with ICS in the previous two months.
* Have a PC20 methacholine less than 8 mg/ml.
* Have a baseline FEV1 greater or equal to 65% of predicted value (at least 6 hours after bronchodilator).
* Are not optimally controlled with short-acting 2 agonists as shown by awakenings due to asthmatic symptoms at least once a week, or regular use of salbutamol on 4 or more occasions per week (excluding exercise prophylaxis) due to asthma symptoms.
* ACQ score equal or greater than 2
* Have sputum eosinophils less than 2%
* Are non smokers or ex-smokers who smoked a maximum of 10 pack/year.

Exclusion Criteria:

* Hospitalized patients within the last 3 months
* Current or recent (within the last month) symptoms of a cold or flu
* Patients with a history of near fatal asthma
* Subjects on inhaled corticosteroids, prednisone, long-acting beta 2 agonists, montelukast or theophylline, within 2 months prior to entry into the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-10; Primary Completion 2010-05 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Lemiere, MD,MSc, Principal Investigator — Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Locations (7):
- Canada (7):
  - Calgary University, Calgary, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Firestone Institute for Respiratory Health, Hamilton, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - The Meakins-Christie Laboratories, Montreal, Quebec
  - Hôpital du Sacré-Coeur de Montréal, Montreal, Quebec
  - Hôpital Laval, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Fluticasone 500 mcg Bid: Treatment with Inhaled Corticosteroids
- Placebo: treatment with placebo
Period: Overall Study
Arm/Group | Fluticasone 500 mcg Bid | Placebo
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluticasone 500 mcg Bid | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (15.3) | 43 (11.7) | 40.5 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 1 | 4 | 5
Region of Enrollment [Number; unit: participants]
  Canada | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Asthma Control Questionnaire (ACQ) Score After 4 Weeks of Treatment With Inhaled Corticosteroids (ICS) or Placebo
Description: Validated questionnaire assessing asthma control after 4 weeks of treatment with ICS or placebo. The ACQ has 7 questions (the top scoring 5 symptoms, FEV1% pred. and daily rescue bronchodilator use). Patients are asked to recall how their asthma has been during the previous week and to respond to the symptom and bronchodilator use questions on a 7-point scale (0=no impairment, 6= maximum impairment). The ACQ score is the mean of 7 items and thus ranges between 0 (well controlled) and 6 (extremely poorly controlled) to yield a mean score out of 6. The higher the score, the worst asthma control is.
Time Frame: Four weeks
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Fluticasone: Treatment with inhaled corticosteroids
- Placebo: Use of placebo inhaler (sham fluticasone)
Arm/Group | Fluticasone | Placebo
Number analyzed (Participants) | 6 | 6
units on a scale | 1.4 (0.5) | 2.2 (0.7)

2. Secondary Outcome: Asthma Quality of Life Questionnaire (AQLQ) Score After 4 Weeks of Treatment
Description: Validated questionnaire assessing quality of life related to asthma after 4 weeks of treatment. The AQLQ is composed of 32 questions in 4 domains (symptoms, activity limitation, emotional function and environmental stimuli). The activity domain contains 5 'patient-specific' questions. This allows patients to select 5 activities in which they are most limited and these activities will be assessed at each follow-up. Patients are asked to think about how they have been during the previous two weeks and to respond to each of the 32 questions on a 7-point scale (7 = not impaired at all - 1 = severely impaired). The AQLQ score is rated on a 7-point scale (1=maximal impairment, 7=no impairment) to yield a mean score out of 7. The worse the quality of life is , the lower the score is.
Time Frame: Four weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fluticasone | Placebo
Number analyzed (Participants) | 6 | 6
units on a scale | 5.5 (1.2) | 4.8 (1.1)

3. Secondary Outcome: Change in Forced Expiratory Volume in One Second (FEV1)
Description: Change in forced expiratory volume in one second (FEV1) after fluticasone or placebo treatment.
Time Frame: Four weeks
Measure: Mean (Standard Deviation); unit: L
Groups:
- Fluticasone: Treatment with Fluticasone
Arm/Group | Fluticasone | Placebo
Number analyzed (Participants) | 6 | 6
L | 0.04 (0.1) | -0.2 (0.2)

4. Secondary Outcome: Change in Provocative Concentration of Methacholine Inducing a 20% Fall in FEV1 (PC20)
Description: Change in provocative concentration of methacholine inducing a 20% fall in FEV1 (PC20) after fluticasone or placebo treatment
Time Frame: Four weeks
Measure: Mean (Standard Deviation); unit: mg/ml
Arm/Group | Fluticasone | Placebo
Number analyzed (Participants) | 6 | 6
mg/ml | 3.4 (0.6) | 2.1 (2.6)

ADVERSE EVENTS:
Arm/Group | Fluticasone 500 mcg Bid | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

LIMITATIONS AND CAVEATS:
Very small sample size. Impossible to recruit the anticipated number of subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No